CLINICAL TRIAL: NCT03007407
Title: A Phase II Study of the Dual Immune Checkpoint Blockade With Durvalumab (MEDI4736) Plus Tremelimumab Following Palliative Hypofractionated Radiation in Patients With Microsatellite Stable (MSS) Metastatic Colorectal Cancer Progressing on Chemotherapy
Brief Title: Study of Durvalumab and Tremelimumab After Radiation for Microsatellite Stable Metastatic Colorectal Cancer Progressing on Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSABP FC-9; ESR-15-11514 (Other: AstraZeneca)
Record Dates: First submitted 2016-12-07; First posted 2017-01-02 (Estimated); Results first posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Cancer Metastatic
Keywords: microsatellite stable; MSS; durvalumab; tremelimumab; mCRC; NSABP
MeSH Terms: interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- durvalumab and tremelimumab (Experimental)
  Interventions: Drug: durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: durvalumab — Following three doses of hypofractionated palliative radiation (Days -2, -1, and Day 0 prior to Cycle 1), patients will receive durvalumab (1500 mg IV infusion) on Day 1 for 4 cycles (in combination with tremelimumab). Beginning with Cycle 5 through Cycle 12, patients will receive durvalumab alone (1500 mg/IV infusion) on Day 1 of each 28 day cycle.
  Other Names: MEDI4736
Drug: Tremelimumab — Following three doses of hypofractionated palliative radiation (Days -2, -1, and Day 0 prior to Cycle 1), patients will receive tremelimumab (75 mg IV infusion) on Day 1 for 4 cycles (in combination with durvalumab).

SUMMARY:
This study is being done to look at the safety and response to the combination of two investigational drugs, tremelimumab and durvalumab, when given after radiation therapy for patients with microsatellite stable (MSS) metastatic colorectal cancer. Tremelimumab and durvalumab recognize specific proteins on the surface of cancer cells and trigger the immune system to destroy the cancer cells.

In order to learn more about certain characteristics of colorectal cancer tumors, this study includes special research tests using samples from diagnostic tumors, fresh tumor samples from an area where the cancer has spread, and blood samples.

DETAILED DESCRIPTION:
The FC-9 study is designed as a phase II, open label, single arm study of the dual immune checkpoint blockade with the combination of durvalumab and tremelimumab following hypofractionated palliative radiation in patients with microsatellite stable (MSS) metastatic colorectal cancer (mCRC) who have progressed on chemotherapy. The primary aim is to determine the anti-tumor efficacy of the dual immune checkpoint blockade with durvalumab plus tremelimumab. The secondary aims are to determine the clinical benefit rate, duration of response, tolerability and correlates of response. Tumor response at unirradiated target lesions will be measured at baseline and every 2 cycles using RECIST 1.1.

Following three doses of hypofractionated palliative radiation (Days -2, -1, and Day 0 prior to Cycle 1), patients will receive the combination of tremelimumab (75 mg IV infusion) and durvalumab (1500 mg IV infusion) on Day 1 for 4 cycles. Beginning with Cycle 5 through Cycle 24, patients will receive durvalumab alone (1500 mg/IV infusion) on Day 1 of each 28 day cycle.

The sample size will be between 12 and 21 evaluable patients. Twelve evaluable patients will be treated in the first stage of the study. If there are no responses among the 12 evaluable patients, the study will be terminated. If the study goes on to the second stage, a total of 21 evaluable patients will be studied.

Submission of tumor tissue and blood samples for FC-9 correlative science studies will be a study requirement for all patients. Requirements will include archived tumor samples from the diagnostic biopsy; additional biopsies of fresh tissue from an accessible lesion prior to radiation therapy and after 2 cycles of study therapy; and blood sample collections.

ELIGIBILITY:
Inclusion Criteria:

* The ECOG performance status must be 0 or 1.
* There must be histologic confirmation of a diagnosis of colorectal adenocarcinoma.
* The tumor must have been determined to be microsatellite stable (MSS).
* There must be documentation by positron emission tomography (PET)/computed tomography (CT) scan, CT scan, or magnetic resonance imaging (MRI), that the patient has evidence of measurable metastatic disease per RECIST 1.1.
* Patients must have an accessible metastatic lesion for pretreatment core biopsy.
* Unless either drug is medically contraindicated, patients must have received oxaliplatin and irinotecan as part of standard metastatic chemotherapy regimens.
* The patient must have multiple sites of metastatic disease with at least one lesion amenable to treatment with stereotactic radiation therapy (SBRT) in the lung or liver and at least one lesion not being irradiated and meeting RECIST 1.1.
* At the time of study entry, blood counts performed within 2 weeks prior to study entry must meet the following criteria:

  * ANC (absolute neutrophil count) must be greater than or equal to 1500/mm3,
  * Platelet count must be greater than or equal to 100,000/mm3; and
  * Hemoglobin must be greater than or equal to 9 g/dL.
* The following criteria for evidence of adequate hepatic function performed within 2 weeks prior to study entry must be met:

  * Total bilirubin must be less than or equal to 1.5 x ULN (upper limit of normal) for the lab unless the patient has a bilirubin elevation greater than 1.5 x ULN to 3 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin; and
  * AST (aspartate aminotransferase)and ALT (alanine transaminase) must be less than or equal to 2.5 x ULN for the lab with the following exception: for patients with documented liver metastases, AST and ALT must be less than or equal to 5 x ULN.
* Adequate renal function within 4 weeks prior to study entry, defined as serum creatinine less than or equal to 1.5 x ULN for the lab or measured or calculated creatinine clearance greater than 40 mL/min by Cockcroft-Gault formula.
* All hematologic, gastrointestinal, and genitourinary chemotherapy toxicities must be less than Grade 2 at the time study therapy is to begin. (Note: Transfusions may be used to correct hemoglobin for patients experiencing anemia from therapy who otherwise would be eligible for the study.
* Patients with reproductive potential (male/female) must agree to use accepted and highly effective methods of contraception while receiving study therapy and for at least 6 months after the completion of study therapy. The definition of effective method of contraception will be based on the investigator's discretion.
* Female patients must either be of non-reproductive potential (i.e., post-menopausal by history: greater than or equal to 60 years old and no menses for greater than or equal to 1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.

Exclusion Criteria:

* Diagnosis of anal or small bowel carcinoma.
* Colorectal cancer other than adenocarcinoma, e.g., sarcoma, lymphoma, carcinoid.
* Previous therapy with any PD-1 or PD-L1 (programmed cell death-1 (PD-1) protein, programmed death ligand-1 (PDL-1) protein inhibitor including durvalumab or anti-CTLA4 (including tremelimumab) for any malignancy.
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving study therapy.
* Active or chronic hepatitis B or hepatitis C.
* Symptomatic or uncontrolled brain metastases requiring concurrent treatments, uncontrolled spinal cord compression, carcinomatous meningitis, or new evidence of brain or leptomeningeal disease; uncontrolled seizures.
* Active infection or chronic infection requiring chronic suppressive antibiotics.
* Active or documented inflammatory disease.
* Known history of human immunodeficiency virus (HIV) or acquired immunodeficiency-related (AIDS) illnesses.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of study therapy with the exceptions of intranasal corticosteroids or systemic corticosteroids at physiological doses that do not exceed 10mg/day of prednisone or an equivalent corticosteroid.
* History of allogeneic organ transplantation.
* Any of the following cardiac conditions:

  * Documented NYHA (New York Heart Association) Class III or IV congestive heart failure,
  * Myocardial infarction within 6 months prior to study entry,
  * Unstable angina within 6 months prior to study entry,
  * Symptomatic arrhythmia. If QTc (corrected QT interval) greater than or equal to 470ms, confirmation of eligible QTc requires mean calculation from 2 additional electrocardiograms (ECGs) 2-5 minutes apart using Fridericia's Correction Formula (mean less than 470 ms).
* Uncontrolled high blood pressure defined as systolic blood pressure (BP) greater than or equal to 150 mmHg or diastolic BP greater than or equal to 100 mmHg with or without anti-hypertensive medication. Patients with initial BP elevations are eligible if initiation or adjustment of BP medication lowers pressure to meet entry criteria.
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* Ongoing or active gastritis or peptic ulcer disease.
* Active bleeding diatheses.
* Known history of previous diagnosis of tuberculosis.
* History of hypersensitivity to durvalumab or tremelimumab or any excipients of these drugs.
* Known history or confirmation of active pneumonia, pneumonitis, symptomatic interstitial lung disease, or definitive evidence of interstitial lung disease described on CT scan, MRI, or chest x-ray in asymptomatic patients; dyspnea at rest requiring current continuous oxygen therapy.
* Active or prior documented autoimmune disease within the past 2 years. (Note: Patients with vitiligo, Grave disease, or psoriasis not requiring systemic treatment within the past 2 years are eligible.)
* Other malignancies unless the patient is considered to be disease-free and has completed therapy for the malignancy greater than or equal to 12 months prior to study entry. Patients with the following cancers are eligible if diagnosed and treated within the past 12 months: carcinoma in situ of the cervix, and basal cell and squamous cell carcinoma of the skin.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements or interfere with interpretation of study results.
* Pregnancy or lactation at the time of study entry. (Note: Pregnancy testing should be performed within 14 days prior to study entry according to institutional standards for women of childbearing potential.)
* Use of any investigational agent. Use and/or receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal anti-bodies) within 14 days prior to the first dose of study therapy.
* Use of any investigational agent within 4 weeks of starting study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (18):
- United States (18):
  - City of Hope, Duarte, California
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center at North Haven, North Haven, Connecticut
  - UF Health Davis Cancer Pavilion and Shands Med Plaza, Gainesville, Florida
  - UF Health Shands Cancer Hospital, Gainesville, Florida
  - UF Health Shands Hospital, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - University of Florida Health Cancer Center at Orlando Health, Orlando, Florida
  - Centralia Oncology Clinic, Centralia, Illinois
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Cancer Care Specialists of Central Illinois/Crossroads Cancer Center, Effingham, Illinois
  - Cancer Care Specialists of Central Illinois-Swansea, Swansea, Illinois
  - Trinity Health Michigan, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - St. Joseph Mercy-Brighton, Brighton, Michigan
  - St. Joseph Mercy-Canton, Canton, Michigan
  - St Joseph Mercy-Chelsea, Chelsea, Michigan
  - Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Durvalumab and Tremelimumab
Started | 33
Completed | 21
Not Completed | 12

BASELINE CHARACTERISTICS:
Population: Participant could identify as more than one race/ethnicity and may be counted in more than one race/ethnicity category.
Arm/Group | Durvalumab and Tremelimumab
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 58 [37 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  Black | 1
  White | 18
  Non Hispanic | 21

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response Rate (ORR) of Dual Immune Checkpoint Blockade by RECIST 1.1
Description: Complete Response (CR): Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be <10mm on the short axis.
  Partial Response (PR): 30% or more decrease in the sum of diameters of target lesions. The reference the baseline sums of diameters. Progressive Disease (PD): 20% or more increase in the sum of diameters of target lesions. The reference is the smallest sum while on study (including the baseline sum if that is the smallest on study). In addition to the relative 20% increase, the sum must also demonstrate an absolute increase 5mm or more. (Note: any appearance of one or more new lesions is also considered progression).Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. The reference is the smallest sum of diameters while on study.
Time Frame: Through treatment, up to 1.3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab and Tremelimumab
Number analyzed (Participants) | 21
percentage of participants | 9.52 [1.17 to 30.38]

2. Secondary Outcome: Percentage of Patients Who Have Achieved Clinical Benefit
Description: Percentage of patients who have achieved clinical benefit defined as CR (complete response) and PR (partial response) and stable disease that lasts at least 4 months
Time Frame: At 16 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab and Tremelimumab
Number analyzed (Participants) | 21
percentage of participants | 14.29 [3.05 to 36.34]

3. Secondary Outcome: Median Duration of Response to mCRC (Metastic Colorectal Cancer) Responds to Study Therapy
Description: Median time from study entry until documentation of progression (years) in half of the patients as determined by RECIST 1.1.
Time Frame: Through study completetion (1.3 years)
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Durvalumab and Tremelimumab
Number analyzed (Participants) | 21
years | 0.85 [0 to NA] — The upper limit of the 95% CI is infinite.

4. Secondary Outcome: Frequency of Adverse Events Assessed by CTCAE 4.0, From Beginning of Treatment to 90 Days After Last Dose
Description: Frequency of adverse events categorized using the NCI Common Terminology Criteria for Adverse Events version 4.0
Time Frame: During treatment (max of 12 cycles; each cycle 28 days) to 90 days after last dose of study therapy
Population: Number of participants analyzed represents the number of patients with toxicity information (29).
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab and Tremelimumab
Number analyzed (Participants) | 29
Participants
  Total | 29
  Grade 0 | 2
  Grade 1 | 3
  Grade 2 | 6
  Grade 3 | 14
  Grade 4 | 3
  Grade 5 | 1

ADVERSE EVENTS:
Time Frame: From the first dose of study therapy until 90 days after the last dose of study therapy.
Arm/Group | Durvalumab and Tremelimumab
All-Cause Mortality (participants affected / at risk) | 6/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 29/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Durvalumab and Tremelimumab (N=29)
Anemia (Blood and lymphatic system disorders) | 3
Hypothyroidism (Endocrine disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 11
Fever (General disorders) | 5
Non-cardiac chest pain (General disorders) | 2
Weight loss (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 2
Itching (Skin and subcutaneous tissue disorders) | 3
Maculopapular rash (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT03007407/Prot_SAP_000.pdf